CLINICAL TRIAL: NCT03437941
Title: Phase 1/2a Dose-Escalation and Expansion Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of CORT125281 With Enzalutamide in Patients With Metastatic Castration-Resistant Prostate Cancer
Brief Title: Study to Evaluate CORT125281 in Combination With Enzalutamide in Patients With mCRPC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CORT125281-601
Record Dates: First submitted 2018-01-16; First posted 2018-02-19 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer
Keywords: Prostate Cancer; Castration-Resistant Prostate Cancer; Glucocorticoid receptor; Antagonist; mCRPC; enzalutamide; androgen receptor
MeSH Terms: conditions — Prostatic Neoplasms; Bulbo-Spinal Atrophy, X-Linked | interventions — enzalutamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Dose Determination Segment 1 (Experimental): Patients will be treated with enzalutamide monotherapy once daily for 28 days followed by combination treatment with CORT125281 at escalating dose levels and enzalutamide once daily in 28-day dosing cycles.
  Interventions: Drug: CORT125281; Drug: Enzalutamide (Xtandi)
- Dose Expansion - Abi-Resistant Cohort (Experimental): Patients who have progressed during treatment with abiraterone and no other AR-blocking therapies will be treated with CORT125281 and enzalutamide.
  Interventions: Drug: CORT125281; Drug: Enzalutamide (Xtandi)
- Dose Expansion - Abi-Resistant Cohort Food Effect (Experimental): Sub-Cohort (first 10 patients enrolled into Cohort A). Patients enrolled into this subcohort will receive a single dose of CORT125281 at Cycle 1 Day -7 and a single dose of CORT125281 at Cycle 1 Day 1 30 minutes after a standard breakfast to assess the effect of food on PK parameters. Patients will then begin CORT125281 in combination with enzalutamide on Cycle 1 Day 2 and continue in 28-day dosing cycles.
  Interventions: Drug: CORT125281; Drug: Enzalutamide (Xtandi)
- Dose Expansion - ARant-Resistant Cohort (Experimental): Patients who progressed during treatment with enzalutamide or second-generation AR-blocking therapies will be treated with a daily dose of CORT125281 and enzalutamide.
  Interventions: Drug: CORT125281; Drug: Enzalutamide (Xtandi)
- Dose Determination Segment 2 (Double-Blind) - Arm A (Experimental): Patients randomized to this cohort will receive enzalutamide and a titrated dose of CORT125281. Enzalutamide will be continued at the dose currently tolerated by the patient at screening.
  Interventions: Drug: CORT125281; Drug: Enzalutamide (Xtandi)
- Dose Determination Segment 2 (Double-Blind) - Arm B (Experimental): Patients randomized to this cohort will receive enzalutamide, placebo, and CORT125281.
  Interventions: Drug: CORT125281; Drug: Enzalutamide (Xtandi); Drug: Placebo

INTERVENTIONS:
Drug: CORT125281 — CORT125281 is supplied as capsules for oral dosing
Drug: Enzalutamide (Xtandi) — Enzalutamide will be taken orally
Drug: Placebo — Placebo capsules to match the appearance of the CORT125281
  Arms: Dose Determination Segment 2 (Double-Blind) - Arm B

SUMMARY:
This is an open-label, Phase 1/2a dose escalation study with an expansion phase to evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD), and preliminary efficacy of CORT125281 in combination with enzalutamide in patients with metastatic castration-resistant prostate cancer (mCRPC) to identify a recommended dose (RD) for Phase 2 studies.

DETAILED DESCRIPTION:
CORT125281 is a selective glucocorticoid receptor (GR) antagonist. In this study, CORT125281 will be administered orally in combination with enzalutamide to patients with metastatic castration-resistant prostate cancer (mCRPC) to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary efficacy of the regimen. The study consists of two phases: a dose-determination phase and an expansion phase. The dose determination phase is designed to determine dose-limiting toxicities and the RD of CORT125281 plus enzalutamide in patients with mCRPC. Once the recommended dosing regimen has been determined, the following expansion cohorts will be enrolled and treated with CORT125281 plus enzalutamide at the recommended dose level.

Abi-Resistant Cohort: Patients who have progressed during treatment with abiraterone, and have received no other androgen receptor (AR)-blocking therapies

ARant-Resistant Cohort: Patients who have progressed during treatment with enzalutamide or other second-generation AR inhibitors.

The effect of food on CORT125281 PK will be assessed in a portion of the patients enrolled in the Expansion Phase. The two expansion cohorts will be enrolled in parallel.

In each phase of the study, routine assessments of safety and tolerability will be performed and samples will be collected to determine standard PK parameters for CORT125281, enzalutamide, and their major metabolites. PD, quality of life evaluations and preliminary evaluations of anti-tumor activity of CORT125281 with enzalutamide will be performed throughout the study.

ELIGIBILITY:
Major Inclusion Criteria:

* Able to understand the purpose and risks of the study; willing and able to adhere to scheduled visits, treatment plans, laboratory tests, and other study evaluations and procedures, and provide written informed consent
* Males ≥18 years of age at the time of signing consent
* Histologically confirmed adenocarcinoma of the prostate with metastatic disease
* Dose-Determination Phase Segment 1 and Expansion Phase: Progressive disease as defined by PSA or imaging after most recent prior therapy. PSA ≥1 ng/mL, if a confirmed rise in PSA is the only indication of progression. Progression by PSA requires rising PSA over a previous reference value by at least 2 measurements obtained ≥1 week apart. PSA measurements can be collected during or after the most recent prior therapy.
* Dose-Determination Phase Segment 2: Currently receiving enzalutamide with a rising PSA as follows:

  1. Rising PSA: 25% increase over nadir and an absolute value of >1 ng/mL by at least 2 measurements obtained ≥1 week apart. PSA measurements can be collected during or after the most recent prior therapy.
  2. Patients must have received enzalutamide for a minimum of 12 weeks and be on stable doses of enzalutamide ≥80 mg QD for at least 4 weeks prior to Cycle 1 Day 1. Patients will continue enzalutamide without interruption during the Screening Period (no wash-out period). This will be the enzalutamide starting dose for combination with CORT125281 beginning on Cycle 1 Day 1.
  3. M0 disease is allowed
* Expansion Phase: Patients must have progressed while receiving an androgen-directed therapy as follows:

  1. Abi-Resistant Cohort: Patients must have progressed during treatment with abiraterone.
  2. ARant-Resistant Cohort: Patients must have progressed during treatment with enzalutamide or second-generation AR-blocking therapies. Patients progressing on enzalutamide immediately prior to enrolling in this study must be on stable doses of enzalutamide. These patients will continue enzalutamide without interruption during the Screening Period (no wash-out period required).
* Baseline tumor assessment performed within 28 days prior to the first dose of study treatment (CORT125281 and/or on-study enzalutamide, whichever is earliest)
* Prior surgical or chemical castration with serum testosterone <1.7 nmol/L (50 ng/dL). If the method of castration is use of a luteinizing hormone releasing hormone (LHRH) analogue,there must be a plan to maintain effective LHRH analogue treatment for the duration of the trial
* Consent to have all protocol required pharmacodynamic biomarker samples, including the pretreatment and on treatment paired tumor biopsies (mandatory for a subset of patients).
* Consent to provide mandatory pharmacogenomic blood sample (Dose-Determination Segment 1 only)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate baseline organ function within 14 days prior to the first dose of study treatment (on-study enzalutamide and/or CORT125281, whichever is earliest)
* Patients receiving systemic corticosteroids greater than 2-weeks in duration within 3 months of study entry or with clinical evidence of adrenal insufficiency must have evidence of adequate adrenal function based upon morning plasma cortisol concentration or ACTH (cosyntropin) stimulation test
* If a patient engages in sexual intercourse with a woman of childbearing potential, a condom with spermicide and another form of birth control must be used during and for 100 days after the final dose of study treatment (CORT125281 or enzalutamide, whichever is latest). A condom is required during and for 100 days after completing treatment with enzalutamide if a patient is engaged in sexual activity with a pregnant woman. Patients must also agree to avoid sperm donation during the study and for at least 100 days after the final treatment administration.

Major Exclusion Criteria:

* Received chemotherapy, non-palliative radiotherapy, immunotherapy, or any investigational cancer therapies within 21 days prior to the first dose of CORT125281, or treatment with such therapies is planned during protocol treatment. Concomitant anticancer therapy is not permitted during the enzalutamide Lead-in Period during Dose-Determination Phase Segment 1
* More than two prior cytotoxic chemotherapy regimens for the treatment of mCRPC

Dose Determination Phase and Expansion Phases will exclude patients for the following:

* Dose-Determination Phase (Segment 1 only)
* Progressed during treatment with enzalutamide prior to Cycle 1 Day -28 (only applies to patients receiving enzalutamide Lead-in) or
* Received prior 2nd generation anti-androgen and require urgent disease response or stabilization
* Expansion Phase Abi-Resistant Cohort:

  * Received prior treatment with enzalutamide, or
  * Received prior 2nd generation anti-androgen and require urgent disease response or stabilization
* Expansion Phase ARant-Resistant Cohort: Require urgent disease response or stabilization
* Ongoing or anticipated therapy with hormone therapy (other than LHRH analogue), including any dose of megestrol acetate (Megace), finasteride (Proscar), dutasteride (Avodart) or received abiraterone within 28 days prior to the first dose of CORT125281
* Contraindication or precaution for enzalutamide
* Parenchymal brain metastases
* Any clinically significant uncontrolled condition that may increase the risk to the study patient or that the Investigator considers places the patient at unacceptable risk
* Received herbal products or alternative therapies that may decrease PSA levels or that may have hormonal anti-prostate cancer activity (e.g., saw palmetto, PC-SPES, PC- HOPE, St. John's wort, selenium supplements, grape seed extract, etc.) within 28 days of study treatment initiation or plans to initiate treatment with these products/alternative therapies during the entire duration of the study
* Received systemic glucocorticoids within 21 days prior to the first dose of CORT125281, or requirement for chronic or frequently used systemic or inhaled glucocorticoids for medical conditions (e.g., rheumatoid arthritis, immunosuppression after organ transplantation). Short courses (<5 days) for non-cancer related reasons are allowed if clinically required (such as prophylaxis for CT).
* Concurrent therapy with strong inhibitors or inducers of CYP3A4 or CYP2C8 or with sensitive substrates of CYP3A4, CYP2C9 or CYP2C19

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only patients with histologically confirmed metastatic castration-resistant prostate cancer will be considered for the study.
Enrollment: 39 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 10 months
  Determine the maximum tolerated dose (MTD) and/or biologically active doses of CORT125281 in combination with enzalutamide to identify the recommended dose (RD) for Phase 2 studies based on the number of patients with dose limiting toxicities (DLTs) of CORT125281 in combination with enzalutamide

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 24 months
  The safety of each treatment group will be assessed by evaluating the incidence of treatment-related adverse events according to CTCAE v4.03
AUC 0-last Pharmacokinetic (PK) parameter | Cycle 1 Day 1 through Cycle 3 Day 1
  Area under the plasma concentration-time curve calculated using linear trapezoidal summation from time 0 to time last, where "last" is the time of the last measurable concentration
AUC 0-24hr PK parameter | Cycle 1 Day 1 through Cycle 3 Day 1
  Area under the plasma concentration-time curve from 0 to 24 hours, calculated using linear trapezoidal summation
AUC 0-infinity PK parameter | Cycle 1 Day 1 through Cycle 3 Day 1
  Area under the plasma concentration-time curve from 0 to infinity, calculated using the formula: AUC0-ing = AUC0-last + Clast/ λz, where λz is the apparent terminal elimination rate constant (whenever possible)
Cmax PK parameter | Cycle 1 Day 1 through Cycle 3 Day 1
  Maximum observed plasma concentration
Cmin,ss PK parameter | Cycle 1 Day 1 through Cycle 3 Day 1
  Minimum observed plasma concentration, at predose at steady-state
CL/F PK parameter | Cycle 1 Day 1 through Cycle 3 Day 1
  Apparent oral clearance
Tmax PK parameter | Cycle 1 Day 1 through Cycle 3 Day 1
  Time of the maximum plasma concentration (obtained without interpolation)
λz PK parameter | Cycle 1 Day 1 through Cycle 3 Day 1
  Terminal elimination rate constant (whenever possible)
Effect of food on the Cmax PK of CORT125281 | Cycle 1 Day -7
  Comparison of the fed state versus the fasted state comparison for the maximum observed plasma concentration (Cmax)
Effect of food on the AUC0-t PK of CORT125281 | Cycle 1 Day -7
  Comparison of the fed state versus fasted state comparison for area under the plasma concentration-time curve
Effect of food on the AUCinf PK of CORT125281 | Cycle 1 Day -7
  Comparison of the fed state versus fasted state comparison for area under the plasma concentration-time curve to infinity
Objective Response Rate (ORR) | 12 months from the enrollment of the final subject
  Determine the ORR by comparing the proportion of the patients who have either a complete response (CR) or partial response (PR)
Reduction in prostate-specific antigen (PSA) | 12 months from the enrollment of the final subject
  Determine the proportion of patients with a reduction in PSA level by >50%
Time to symptomatic skeletal event (SSE) | 12 months from the enrollment of the final subject
  Determine the time to SSE defined as symptomatic fracture, radiation or surgery to bone, or spinal cord compression
Radiographic progression-free survival (rPFS) | Baseline to 12 months
  Determine rPFS defined as the time interval from first dose of study drug (CORT125281 and/or enzalutamide) to the date when the first site of disease is found to progress on CT, MRI, or radionucleotide bone scan per PCWG3, or death whichever occurs first; including the proportion of patients progression-free at 4, 6, and 12 months
Time to prostate-specific antigen (PSA) progression | Baseline to 12 months
  Assess time to PSA progression, including the proportion of patients progression free at 4, 6, and 12 months
Time to clinical progression | Baseline to 12 months
  Assess time to clinical progression, including the proportion of patients progression free at 4, 6, and 12 months
Duration of Response (DOR) | 12 months from the enrollment of the final subject
  Determine the DOR by the time from the first occurrence of a documented objective tumor response to the time of radiographic progression (per investigator using RECIST v1.1) or death from any cause on study, whichever occurs first
Overall Survival (OS) | 12 months from the enrollment of the final subject
  Determine OS by the time from the first dose of study drug (CORT125281 and/or enzalutamide) to the date of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: William Guyer, PharmD, Study Director — Corcept Therapeutics; Grace Mann, PhD, Study Director — Corcept Therapeutics
Locations (8):
- United States (5):
  - Scottsdale, Scottsdale, Arizona
  - Detroit, Detroit, Michigan
  - New York, New York, New York
  - Portland, Portland, Oregon
  - Madison, Madison, Wisconsin
- United Kingdom (3):
  - London, London, England
  - Southampton, Southampton, England
  - Sutton, Sutton, Surrey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Serritella AV, Shevrin D, Heath EI, Wade JL, Martinez E, Anderson A, Schonhoft J, Chu YL, Karrison T, Stadler WM, Szmulewitz RZ. Phase I/II Trial of Enzalutamide and Mifepristone, a Glucocorticoid Receptor Antagonist, for Metastatic Castration-Resistant Prostate Cancer. Clin Cancer Res. 2022 Apr 14;28(8):1549-1559. doi: 10.1158/1078-0432.CCR-21-4049. PMID 35110415